CLINICAL TRIAL: NCT02386813
Title: International Extranodal NK/T-cell Lymphoma Project: Prognostic Factors in the Era of Nonanthracycline-based Treatment
Brief Title: International Extranodal NK/T-cell Lymphoma Project
Acronym: PINK
Status: Completed | Type: Observational
Sponsor: Samsung Medical Center (Other)
Collaborators: Seok Jin Kim (Unknown); Consortium for Improving Survival of Lymphoma (Other); Asia Lymphoma Study Group (Unknown); Lymphoma Study Association (Other); Dok Hyun Yoon (Unknown); Arnaud Jaccard (Unknown); Wee Joo Chng (Unknown); Soon Thye Lim (Unknown); Huangming Hong (Unknown); Yong Park (Unknown); Kian Meng Chang (Unknown); Yoshinobu Maeda (Unknown); Fumihiro Ishida (Unknown); Dong-Yeop Shin (Unknown); Jin Seok Kim (Unknown); Seong Hyun Jeong (Unknown); Deok-Hwan Yang (Unknown); Jae-Cheol Jo (Unknown); Gyeong-Won Lee (Unknown); Chul Won Choi (Unknown); Won-Sik Lee (Unknown); Tsai-Yun Chen (Unknown); Kiyeun Kim (Unknown); Sin-Ho Jung (Unknown); Tohru Murayama (Unknown); Yasuhiro Oki (Unknown); Ranjana Advani (Unknown); Francesco d'Amore (Unknown); Norbert Schmitz (Unknown); Cheolwon Suh (Unknown); Ritsuro Suzuki (Unknown); Yok Lam Kwong (Unknown); Tong-Yu Lin (Unknown)
Responsible Party: Principal Investigator, Won Seog Kim, Professor, Samsung Medical Center
Other Study IDs: 2013-03-071
Record Dates: First submitted 2015-03-06; First posted 2015-03-12 (Estimated); Last update posted 2017-04-11 (Actual); Status verified 2017-04

CONDITIONS: Extranodal NK/T-cell Lymphoma, Nasal Type
MeSH Terms: conditions — Lymphoma, Extranodal NK-T-Cell

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Training cohort: 1. Patients diagnosed with ENKTL, nasal type between January 1, 1995 and December 31, 2013;
  2. Patients treated with non-anthracycline based therapy as an initial treatment.
- Validation cohort: 1. Patients diagnosed with ENKTL, nasal type between January 1, 1998 and December 31, 2014;
  2. Patients treated with non-anthracycline based therapy as an initial treatment.

SUMMARY:
This study is to explore risk factors for poor progression-free survival (PFS) and overall survival (OS) in ENKTL, and establish a prognostic model for ENKTL patients treated with non-anthracycline based treatment.

DETAILED DESCRIPTION:
This is a retrospective cohort study using anonymized information from patients with ENKTL. The following criteria are required: (1) Patients diagnosed with ENKTL, nasal type between January 1, 1995 and December 31, 2014; (2) Patients treated with non-anthracycline based therapy as an initial treatment. The pathology of initial diagnosis was reviewed by designated pathologists.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with ENKTL, nasal type
* Patients diagnosed between January 1, 1995 and December 31, 2014
* Patients treated with nonanthracycline-based therapy as the initial treatment after diagnosis
* Nonanthracycline-based therapy includes the following treatments:
* Radiotherapy including concurrent chemoradiation
* Chemotherapy not including anthracycline such as doxorubicin (e.g. SMILE, VIPD) The type of salvage treatment will not be a criterion for exclusion. Thus, patients who had received various kinds of salvage treatment including anthracycline-containing regimens can be included. Patients who had undergone autologous or allogeneic stem cell transplantation can also be included in the analysis if they satisfy the above-mentioned inclusion criteria.

Exclusion Criteria:

* Patients who had received anthracycline-based therapy, such as CHOP or CHOP-like regimens, as the initial treatment.
* Patients who do not have pathology slides available for central review.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: 1. Patients diagnosed with ENKTL, nasal type between January 1, 1995 and December 31, 2014;
  2. Patients treated with non-anthracycline based therapy as an initial treatment.
Sampling Method: Probability Sample
Enrollment: 770 (Actual)
Dates: Start 2013-01; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Overall survival | 5 year
  Time between the date of diagnosis and any kinds of death

SECONDARY OUTCOMES:
Progression-free survival | 5 year
  Time between the date of diagnosis and any kinds of death or relapse/progression

CONTACTS AND LOCATIONS:
Overall Officials: Won Seog Kim, MD, PhD, Principal Investigator — Samsung Medical Center
Locations (1):
- Samsung Medical Center, Seoul, South Korea